CLINICAL TRIAL: NCT07255586
Title: Self-monitoring of Hearing Aids Using Artificial Intelligence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sodra Alvsborgs Hospital (Other)
Responsible Party: Principal Investigator, Milijana Malmberg, Principal Investigator, Sodra Alvsborgs Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Self-monitoring of HAs
Record Dates: First submitted 2025-09-30; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Self-monitoring of hearing aids. ALl participants in this group are offered self-monitoring of hearing aids.
  Interventions: Device: Self-monitoring of hearing aids using artificial intelligence
- Standard care (Other): All participants in this group are offered traditional hearing care.
  Interventions: Other: Traditional hearing care at our clinics.

INTERVENTIONS:
Device: Self-monitoring of hearing aids using artificial intelligence — Self-monitoring of hearing aids using artificial intelligence
  Arms: Intervention group
Other: Traditional hearing care at our clinics. — Traditional hearing care at our clinics
  Arms: Standard care

SUMMARY:
This project investigates how self-monitoring of hearing aids through an AI-based mobile app can complement physical and digital healthcare visits. The aim is to increase patient involvement in rehabilitation, enable hearing aid adjustments in everyday sound environments, and improve access to hearing care.

DETAILED DESCRIPTION:
Considering the growing population, healthcare is increasingly focusing on integrating digital solutions into care. Such solutions typically require active patient participation and have the potential to positively impact person-centered care.

The purpose of this project is to investigate the outcomes of complementing physical and/or digital hearing care visits with patient self-monitoring of hearing aids. Participants will undergo the standard steps of the hearing rehabilitation process. In addition, the intervention group will be offered the opportunity to self-monitor their hearing aids between physical and/or digital appointments using artificial intelligence (AI) integrated into a mobile application provided by a hearing aid supplier.

The focus is to increase patient involvement in the rehabilitation process, utilize adjustment possibilities in everyday sound environments, and improve access to hearing care for the target population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are eligible for a new or renewed hearing rehabilitation process at four of the Hearing organizations audiology clinics

Exclusion Criteria:

* Not fullfilling the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Hearing Handicap Inventory for the Elderly-Screening | From enrollment to the end of treatment at 6 months
  Evaluates self-perceived psychosocial and emotional effects of hearing loss. Min 0 to max 100 points. Higher points equal greater self-perceived hearing problems.

SECONDARY OUTCOMES:
Client Oriented Scale of Improvement | From enrollment to the end of treatment at 6 months
  Not reporting score on a scale.
Communication Strategies Scale of the Communication Profile for the Hearing Impaired | From enrollment to the end of treatment at 6 months
  The CSS includes three subscales: the Maladaptive Behaviours, nine questions addressing strategies that complicate communication, and Verbal Strategies and Nonverbal Strategies, both of which address 16 items related to strategies that can improve communication. The scoring for all three subscales reflects how frequently a specific strategy occurs in different situations.

OTHER OUTCOMES:
International Outcome Inventory for Hearing Aids | At the end of treatment at 6 months
  The IOI-HA measures seven different variables where higher points equal better outcomes. The variables are use, benefit, activity limitation, satisfaction, participation restriction, impact on environment, and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Milijana M Malmberg, PhD, Principal Investigator — Habilitering & Hälsa

IPD SHARING:
Plan to Share IPD: No